CLINICAL TRIAL: NCT01261572
Title: ASP3550 Phase II Study - A Maintenance-Dose-Finding Study of Three-Month Depot in Patients With Prostate Cancer -
Brief Title: Study to Find Maintenance Dose for Periodic Administration of ASP3550
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3550-CL-0009
Record Dates: First submitted 2010-12-01; First posted 2010-12-16 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Degarelix; ASP3550; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose group (Experimental): ASP3350 high dose
  Interventions: Drug: degarelix
- Low dose group (Experimental): ASP3350 low dose
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix — periodic injection
  Other Names: ASP3550

SUMMARY:
To find effective doses of ASP3550 on the maintenance of serum testosterone suppression in patients with prostate cancer.

DETAILED DESCRIPTION:
ASP3550 is administered periodically to patients with prostate cancer. The primary efficacy variable is the effect of ASP3550 on the maintenance of serum testosterone suppression. In addition, the safety and pharmacokinetics of ASP3550 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer (adenocarcinoma) of all stages
* A patient in whom endocrine treatment is indicated. Patients with rising serum PSA after having prostatectomy or radiotherapy performed with curative intention
* Serum testosterone level above 2.2 ng/mL
* An ECOG (Eastern Co-operative Oncology Group) P.S. (Performance Status) score of 0 to 2
* Serum PSA level above 2 ng/mL

Exclusion Criteria:

* Previous or present endocrine treatment for prostate cancer.

However, patients who have undergone neoadjuvant/adjuvant endocrine therapy for a maximal duration of 6 months and in whom prostatectomy or radiotherapy was terminated at least 6 months

* Treated with a 5α-reductase inhibitor
* A candidate for curative therapy, i.e., radical prostatectomy or radiotherapy within 12 months
* Concurrent or a history of severe liver disease
* Abnormal ECG such as long QTc
* A patient receiving ASP3550 in past times
* Administered drug in another clinical study or a post-market clinical study in the 28 days prior to the study

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-10-12 (Actual); Primary Completion 2012-04-24 (Actual); Study Completion 2012-04-24 (Actual)

PRIMARY OUTCOMES:
Change in proportion of patients with serum testosterone ≤0.5 ng/mL over time | Baseline and for one year

SECONDARY OUTCOMES:
Changes in serum level of testosterone over time | Baseline and for one year
Changes in serum level of Luteinizing Hormone (LH) over time | Baseline and for one year
Changes in serum level of Follicle Stimulating Hormone (FSH) over time | Baseline and for one year
Changes in serum level of Prostate Specific Antigen (PSA) over time | Baseline and for one year
Time to the recurrence of serum PSA | For one year
Safety evaluated by the incidence of Adverse Events (AEs), physical exam and results of lab tests | One year

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shuku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=311